CLINICAL TRIAL: NCT06322264
Title: Promoting Children's Participation in Conventional X-ray Examinations
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-05435-01
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Heart Rate Determination; Patient Participation
Keywords: Children's participation; Conventional x-ray procedure; Variation in heart rate
MeSH Terms: conditions — Patient Participation | interventions — Heart Rate

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric patients: Pediatric patients between the ages of 4 and 12 undergoing conventional X-ray examinations.
  Interventions: Diagnostic Test: Measurement of variation in heart rate
- Parents: Parents of the included pediatric patients between the ages of 4 and 12 undergoing conventional X-ray examinations.
- Radiographers: Radiographers who examine the included pediatric patients between the ages of 4 and 12 undergoing conventional X-ray examinations.

INTERVENTIONS:
Diagnostic Test: Measurement of variation in heart rate — The children will be given a portable device that will monitor their heart rate, enabling the recording of the rate of their pulse.
  Groups: Pediatric patients

SUMMARY:
The goal of this explorative observational study is to map the procedure and child centered approach in the examination for children that undergo conventional X-ray examinations. The main questions aim to answer:

* How many images need to be retaken during conventional X-ray examinations?
* What is the reason why the pictures need to be redone?
* What is the time required for the various examinations?
* What experience of the procedure of the examination is there among those involved?
* Can the physical impact be observed through variation in heart rate in children that undergo conventional X-ray examinations?

Participants will answer questionnaires about the children's participation in the procedure and the variation in heart rate will be measured on the children who undergo the examinations.

DETAILED DESCRIPTION:
Many children receive healthcare services during their childhood. In Sweden, approximately 330,000 children aged 0-15 require conventional X-ray examinations annually. It is imperative that the justification for conducting these X-ray examinations on children is carefully considered. Improper positioning during the image capturing process can result in inadequate images that do not provide necessary diagnostic information. This may require that the X-ray procedure must be repeated, leading to unnecessary exposure of children to radiation. This situation poses complexities as a means to minimize the occurrence of repeated imaging procedures and minimize unnecessary radiation exposure, children may be subject to some level of restraint.

Effective January 1, 2020, Sweden adopted the United Nations Convention on the Rights of the Child into law, with the aim of enhancing and elucidating the rights of children.

This entails that children are entitled to receive care from personnel who possess the expertise and qualifications necessary to uphold both the physical and mental well-being of children, as well as their rights, prior to, during, and following a procedure such as an X-ray examination.

The radiographer plays a significant role in determining the outcome of pediatric examinations, impacting both the child's experience and the quality of imaging as well as the radiation dose received. This study investigates the perceptions of health care professionals regarding pediatric examinations, focusing on procedure, child centered approach, and overall experience during conventional X-ray procedures. Additionally, it explores the experiences of children and their parents during examinations, including children's level of participation in the process. It is also essential to evaluate the physical indicators, this in the form of changes in the child's pulse rate.

To establish a standard baseline for normal variation, investigators will measure pulse rates before, during, and after an examination using portable heart rate monitors.

The questionnaires will be answered by the population -children, parents and the examining radiographer after each examination has been completed and will mainly consist of shorter multiple-choice options with the possibility of extended answers in cases where additions need to be made.

For the parts that are common between the three groups, the questions to the children are taken from a questionnaire about children's participation. Parents and radiographers receive the same questions and answers on a Likert scale.

A descriptive and comparative analysis will be done with the support of different software, Excel and SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 4-12 yrs who undergo standard x-ray examinations
* parents to the child
* assigned radiographers

Exclusion Criteria:

* Children and parents who have cognitive and/or language difficulties

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population consists of the people who are involved with the child undergoing an X-ray examination.
  Which are the children who are to undergo conventional x-rays and are between the ages of 4-12 years. Those who are accompanying this child and the radiographers who carry out the examination will also be there.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Variation in heart rate | The measurement is done through the examination total time 15 minutes (baseline before start 1-2 minutes, start of exam 2-10 minutes, end of exam after 10-15 minutes)
  To compare the variations in pulse with the experience of the examination

CONTACTS AND LOCATIONS:
Overall Officials: Pether Jildenstål, Assoc. Prof., Study Director — Lund University
Locations (1):
- SUS, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardy M, Armitage G. The child's right to consent to x-ray and imaging investigations: issues of restraint and immobilization from a multidisciplinary perspective. J Child Health Care. 2002 Jun;6(2):107-19. doi: 10.1177/136749350200600204. PMID 12136815
- [Result] Sahlberg S, Karlsson K, Darcy L. Children's rights as law in Sweden-every health-care encounter needs to meet the child's needs. Health Expect. 2020 Aug;23(4):860-869. doi: 10.1111/hex.13060. Epub 2020 Apr 22. PMID 32319716
- [Result] Gilljam BM, Arvidsson S, Nygren JM, Svedberg P. Child participation in health care (ChiPaC)-Development and psychometric evaluation of a self-report instrument for children's participation in health care. J Clin Nurs. 2020 Jan;29(1-2):107-118. doi: 10.1111/jocn.15063. Epub 2019 Oct 10. PMID 31531995
- See also: Almen, A., & Jangland, L., (2020). Radiological examinations in Sweden in 2018 (Report 2020:14). The Radiation Safety Authority. — https://www.stralsakerhetsmyndigheten.se/publikationer/rapporter/stralskydd/2020/202014/